CLINICAL TRIAL: NCT02998593
Title: Effect of Red and White Bahman on Semen Parameters,Testosteron ,LH, FSH and Defragmentation of DNA . A Double Blind Randomised Clinical Trial (Phase 3)
Brief Title: The Effect of Combination of Red and White Bahman Retrieved of Iranian Traditional Medicine on Semen Parameters in Idiopathic Oligospermic Men
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Royan Institute (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Royan-Emb-026
Record Dates: First submitted 2016-11-09; First posted 2016-12-20 (Estimated); Last update posted 2017-04-28 (Actual); Status verified 2016-10

CONDITIONS: Infertility, Male
Keywords: Semen parameters Male infertility oligospermia Traditional Medicine
MeSH Terms: conditions — Infertility, Male

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- extracted red Bahman and white bahman (Experimental): 500 mg of extracted red Bahman and white bahman that is used once a day.
  Interventions: Drug: Bahman capsules
- Placebo (Placebo Comparator): 500 mg of placebo once time a day
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Bahman capsules — Oral Use of Bahman capsules for 3 months by patients.
  Arms: extracted red Bahman and white bahman
Drug: Placebo — Oral use of placebo capsules by patients for 3 months.
  Arms: Placebo

SUMMARY:
This study is a prospective double blind randomized controlled trial to investigate the effect of red and white bahman on semen parameters, sexual hormones and DNA defragmentation in idiopathic oligospermic men .Include patients will take the medicine and placebo in different two case and control groups for 3 month and semen parameters and other variants at the start and end of study.

DETAILED DESCRIPTION:
This is a randomized, double blind; placebo-controlled clinical trial has been started from july 2016 and will continue to july 2016 in Royan institute. The eligible patients who fulfilled the study criteria will be included in the trial.

Study protocol and assays All the patients will have a complete history evaluation and physical examination by the attending urologist who is blinded to the study and enter the study according to inclusion criteria.. semen analysis and hormonal laboratory tests [Testosterone, Luteinizing hormone (LH) Follicle stimulating hormone(FSH)] will done in same lab at start of study and 3 month after. Intervention time is 3 month for each patient. semen analysis wil be done according to who laboratory manual for the examination and processing of human semen 5th edition and hormonal tests (LH,FSH,Testosterone) with Elisa method (with score of International Unit). DNA Defragmentation will evaluate with Sperm Chromatin Structure Assay(SCSA) method. semen parameters which will evaluate is the number of normal and abnormal shape sperms, velocity of sperms, volume and viscosity of semen at start and end of the study. medicine and placebo prescribe in 500mg capsules for 3month. red and white Bahman is an effective medicine in male infertility treatment In Iranian Traditional Medicine. at the end of study main aim of the study is evaluation effect of combination of Red and White Bahman retrieved of Iranian Traditional Medicine on Semen Parameters in Idiopathic Oligospermic . Red Bahman and White bahman ,nutrition ,placebo, smoking and Testosterone,LH,FSH,Concentration,number,sha-pe,of sperm before and after the study is variables of study.

ELIGIBILITY:
Inclusion Criteria:

1. all idiopathic oligospermic patient in range of 20 to 45 years old
2. sperm count under 15 million /ml 3;No history of taking chemical or herbal medicine effective on sperm genesis in last 3 month( like Hormonal drug ,antidepressant ,anti hypertension,cimetidine, cyproteron, sulphasalazine, flutamide, spironolactone, estrogen,opium 4:No history of Varicocele and Obstructive disease 5:;No leukocytospermia

Exclusion Criteria:

Taking chemical or herbal medicine effective on spermatogenesis (hormonal and sperm reducing and increasing agent); 2. ; Increasing BMI > 30 3. Leukocytospermia 4. varicocele

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2016-07; Primary Completion 2017-04 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
Semen analysis | 3 months
  Performing the semen analysis to evaluate the sperm count ,sperm motility and sperm morphology.

SECONDARY OUTCOMES:
Testosterone | 3 months
  Evaluation the testosterone by ELISA level 3 months after intervention.
FSH | 3 months
  Evaluation the FSH level by ELISA 3 months after intervention.
LH | 3 months
  Evaluation the LH level by ELISA 3 months after intervention.
DNA defragmentation | 3 months
  Evaluation the DNA defragmentation by SCSA Method 3 months after intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Hamid Gourabi, PhD, Study Chair — Head of Royan Institute; Seyed Jalil Hosseini, PhD, Study Director — Department of Andrology, Royan Institute for Reproductive Biomedicine, ACECR, Tehran, Iran.; Mahmoudreza Faghihi, MD,PhD, Study Director — Shahid Beheshti University of Medical Science _School of Traditional Medicine,Tehran ,Iran; Mina Movahed, MD,PhD, Principal Investigator — Shahid Beheshti University of Medical Science _School of Traditional Medicine,Tehran ,Iran
Locations (1):
- Royan Institute, Tehran, Iran

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — http://royaninstitute.org